CLINICAL TRIAL: NCT02684006
Title: A PHASE 3, MULTINATIONAL, RANDOMIZED, OPEN-LABEL, PARALLEL-ARM STUDY OF AVELUMAB (MSB0010718C) IN COMBINATION WITH AXITINIB (INLYTA(REGISTERED)) VERSUS SUNITINIB (SUTENT(REGISTERED)) MONOTHERAPY IN THE FIRST-LINE TREATMENT OF PATIENTS WITH ADVANCED RENAL CELL CARCINOMA
Brief Title: A Study of Avelumab With Axitinib Versus Sunitinib In Advanced Renal Cell Cancer (JAVELIN Renal 101)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991003; 2015-002429-20 (EudraCT Number); JAVELIN RENAL 101 (Other: Alias Study Number)
Record Dates: First submitted 2016-01-25; First posted 2016-02-17 (Estimated); Results first posted 2024-10-29 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Renal Cell Cancer
Keywords: Cancer; renal cell cancer; kidney disease; kidney neoplasms; axitinib, sunitinib
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Kidney Diseases; Kidney Neoplasms | interventions — avelumab; Axitinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avelumab in combination with axitinib (Experimental): Avelumab administered at 10 mg/kg IV every two weeks in combination with axitinib, 5 mg PO BID.
  Interventions: Drug: Avelumab (MSB0010718C); Drug: Axitinib (AG-013736)
- Sunitinib (Active Comparator): Sunitinib given at 50 mg PO QD on schedule 4/2
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Avelumab (MSB0010718C) — IV treatment Avelumab administered at 10 mg/kg IV every two weeks
  Arms: Avelumab in combination with axitinib
Drug: Axitinib (AG-013736) — Oral treatment Axitinib given 5 mg PO BID
  Other Names: Inlyta
  Arms: Avelumab in combination with axitinib
Drug: Sunitinib — Oral treatment Sunitinib given at 50 mg PO QD on schedule 4/2
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
This is a phase 3 randomized trial evaluating the anti-tumor activity and safety of avelumab in combination with axitinib and of sunitinib monotherapy, administered as first-line treatment, in patients with advanced renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic RCC with clear cell component
* Availability of a formalin-fixed, paraffin-embedded (FFPE) tumor tissue block from a de novo tumor biopsy during screening (biopsied tumor lesion should not be a RECIST target lesion). Alternatively, a recently obtained archival FFPE tumor tissue block (not cut slides) from a primary or metastatic tumor resection or biopsy can be provided if the following criteria are met: 1) the biopsy or resection was performed within 1 year of randomization AND 2) the patient has not received any intervening systemic anti-cancer treatment from the time the tissue was obtained and randomization onto the current study. If an FFPE tissue block cannot be provided as per documented regulations then, 15 unstained slides (10 minimum) will be acceptable
* Availability of an archival FFPE tumor tissue from primary tumor resection specimen (if not provided per above). If an FFPE tissue block cannot be provided as per documented regulations 15 unstained slides (10 minimum) will be acceptable
* At least one measurable lesion as defined by RECIST version 1.1 that has not been previously irradiated
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow function, renal and liver functions

Exclusion Criteria:

* Prior systemic therapy directed at advanced or metastatic RCC
* Prior adjuvant or neoadjuvant therapy for RCC if disease progression or relapse has occurred during or within 12 months after the last dose of treatment.
* Prior immunotherapy with IL-2, IFN-α, or anti PD 1, anti PD L1, anti PD L2, anti CD137, or anti cytotoxic T lymphocyte associated antigen 4 (CTLA 4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T cell co stimulation or immune checkpoint pathways
* Prior therapy with axitinib and/or sunitinib as well as any prior therapies with other VEGF pathway inhibitors
* Newly diagnosed or active brain metastasis
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3), any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of partially controlled asthma Global Initiative for Asthma 2011)
* Any of the following in the previous 12 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, LVEF less than LLN, clinically significant pericardial effusion, cerebrovascular accident, transient ischemic attack
* Any of the following in the previous 6 months: deep vein thrombosis or symptomatic pulmonary embolism
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza vaccines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 886 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (258):
- United States (90):
  - Southern Cancer Center, Daphne, Alabama
  - Southern Cancer Center, Mobile, Alabama
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - City of Hope National Medical Center, Duarte, California
  - City of Hope, Duarte, California
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC IDS Pharmacy, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Advanced Health Sciences Pavilion, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Cedars-Sinai, Los Angeles, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado Cancer Center Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Hospital - Clinical Trials Office (CTO), Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service- Emory University, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - East Jefferson General Hospital, Metairie, Louisiana
  - East Jefferson Hematology-Oncology Metairie Physician Service Inc., Metairie, Louisiana
  - New England Cancer Specialists, Kennebunk, Maine
  - New England Cancer Specialists, Scarborough, Maine
  - New England Cancer Specialists, Topsham, Maine
  - Oncology Investigational Drug Services- The Sidney Kimmel Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Massachusetts General Hospital Clinical Trials Pharmacy, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center Pharmacy - BIDMC, Boston, Massachusetts
  - Dana - Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Franklin Medical Center, Greenfield, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Barnes-Jewish Hospital, Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, Siteman Cancer Center, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Barnes-Jewish Hospital, Siteman Cancer Center - South County, St Louis, Missouri
  - St. Vincent Healthcare, Billings, Montana
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana, Billings, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - New York Oncology Hematology, PC, Albany, New York
  - New York Oncology Hematology, P.C., Clifton Park, New York
  - Memorial Sloan Kettering Cancer Center - Investigational Drug Service Pharmacy, Long Island City, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYU Investigational Pharmacy, New York, New York
  - NYU Langone Medical Center, New York, New York
  - MSKCC-Monitoring Suite, New York, New York
  - Evelyn H. Lauder Breast and Imaging Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sidney Kimmel Center for Prostate and Urologic Cancers, New York, New York
  - Stony Brook University-Cancer Center, Stony Brook, New York
  - Stony Brook University, Stony Brook, New York
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - The Ohio State University - GU Clinic, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Cancer Care Associates Medical Oncology, Allentown, Pennsylvania
  - St.Luke's Hospital-Allentown Campus, Allentown, Pennsylvania
  - Cancer Care Associate Medical Oncology, Bethlehem, Pennsylvania
  - St. Lukes University Health Network, Bethlehem, Pennsylvania
  - St.Luke's Cancer Center Anderson, Easton, Pennsylvania
  - St.Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Investigational Drug Service, University of Pennsylvania, Philadelphia, Pennsylvania
  - St.Luke's Quakertown Hospital, Quakertown, Pennsylvania
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Gulf Coast, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Investigational Product Center (IPC), Irving, Texas
  - Investigational Products Center (IPC), Irving, Texas
  - Investigational Products Center (lPC), Irving, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Rainier Hematology-Oncology, PC, Puyallup, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Australia (23):
  - Macquarie University Hospital Pharmacy, Macquarie University, New South Wales
  - Macquarie University, Macquarie University, New South Wales
  - Nuclear Medicine Department, Randwick, New South Wales
  - Pharmacy Department, Clinical Trials, Randwick, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Spectrum Medical Imaging, Randwick, New South Wales
  - Division of Cancer Services, Woolloongabba, Queensland
  - BHS Diagnostic Services, Ballarat, Victoria
  - Lake Imaging, Ballarat, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Eastern Health, Box Hill, Victoria
  - Monash Health Translational Precinct, Monash Medical Centre, Clayton, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Monash Cancer Centre, East Bentleigh, Victoria
  - Moorabbin Radiology, East Bentleigh, Victoria
  - Slade Health, Mount Waverley, Victoria
  - Ballarat Day Procedure Centre, Wendouree, Victoria
  - Ballarat Oncology & Haematology Services, Wendouree, Victoria
  - Nova Pharmacy, Wendouree, Victoria
  - SKG Radiology, Murdoch, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God Murdoch Hospital, Murdoch, Western Australia
  - EPIC Pharmacy Murdoch, Perth, Western Australia
- Austria (2):
  - Krankenhaus der Barmherzigen Schwestern Wien, Vienna
  - Medizinische Universitaet Wien, Vienna
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHU de Liège, Liège
- Canada (11):
  - Foothills Medical Centre, Calgary, Alberta
  - Alberta Health Services - Cancer Care, Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Sindi Ahluwalia Hawkins Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - BC Cancer GU Clinic - Fairmont Medical Building, Vancouver, British Columbia
  - London Regional Cancer Program, London Health Sciences Centre, London, Ontario
  - R.S. McLaughlin Durham Regional Cancer Centre, Lakeridge Health, Oshawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CIUSSS de l'Estrie-Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
- Denmark (2):
  - Herlev Hospital, Onkologisk Afdeling R, Herlev
  - Odense Universitetshospital, Odense C
- France (11):
  - Centre Eugene Marquis Service Pharmacie - Essais Cliniques, Rennes, Cedex
  - Centre Francois Baclesse, Caen
  - Centre de Cancérologie de la Sarthe (CCS) - Clinique Victor Hugo, Le Mans
  - Clinique Victor Hugo Centre de Cancerologie de la Sarthe, Le Mans
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Eugene Marquis, Rennes
  - Institut de Cancérologie de l'Ouest - Centre René Gauducheau, Saint-Herblain
  - Institut de Cancerologie de Lorraine (ICL), Vandœuvre-lès-Nancy
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Jena, Jena, Thuringia
  - Universitaetsklinikum Jena Klinik und Poliklinik fuer Urologie, Jena, Thuringia
- Hungary (2):
  - Dél.pesti Centrumkórház-OHII Szent Lálszló Kórház telephely, Budapest
  - Országos Onkológiai Intézet, Budapest
- Israel (10):
  - The Chaim Sheba Medical Center, Tel Litwinsky, Ramat - GAN
  - Assaf Harofe MC, Beer Yaakov
  - Shamir Medical Center, Beer Yaakov
  - Rambam Health Care Campus, Haifa
  - Rambam Healthcare Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Pharmacy - clinical unit, Tel Aviv Sourasky Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Centro di Riferimento Oncologico - IRCCS, Aviano, (PN)
  - Farmacia Studi Clinici, Rozzano, Milan
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - SC Farmacia, Milan
  - Istituto Europeo di Oncologia, Milan
  - Servizio di Farmacia, Milan
  - Azienda Ospedaliera San Camillo Forlanini, Rome
- Japan (16):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University School of Medicine & Hospital, Hirosaki, Aomori
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Akita University Hospital, Akita
  - Chiba Cancer Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - Niigata University Medical & Dental Hospital, Niigata
  - Tokushima University Hospital, Tokushima
  - Yamagata University Hospital, Yamagata
- Mexico (3):
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Centro Universitario Contra el Cancer, Monterrey, Nuevo León
  - Oaxaca Site Management Organization S.C., Oaxaca City
- Netherlands (10):
  - Netherlands Cancer Institute/Antoni van Leeuwenhoek Hospital, Amsterdam, North Holland
  - Netherlands Cancer Institute / Apotheek MC Slotervaart, Amsterdam, North Holland
  - VU University Medical Center (VUmc), Amsterdam, North Holland
  - Sint Franciscus Gasthuis, Pharmacy, Rotterdam, South Holland
  - Sint Franciscus Gasthuis, Rotterdam, South Holland
  - Maxima Medisch Centrum, Eindhoven
  - St Apotheek der Haarlemse Ziekenhuizen, Haarlem
  - Spaarne Gasthuis, Hoofddorp
  - Maastricht University Medical Center, Maastricht
  - Maxima Medisch Centrum, Veldhoven
- New Zealand (11):
  - Auckland City Hospital, Grafton, Auckland
  - Tauranga Hospital, Bay of Plenty Clinical Trials Unit, Tauranga, Bay of Plenty
  - Palmerston North Hospital, Palmerston North, Manawatu-Wanganui
  - Tauranga Hospital, Tauranga Bay of Plenty, Tauranga
  - Wairarapa District Health Board, Masterton, Wairarapa
  - Auckland City Hospital Pharmacy, Auckland
  - Baxter Healthcare New Zealand, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital Pharmacy Services, Hamilton
  - Waikato Hospital, Hamilton
  - Broadway Radiology, Palmerston North
- Romania (4):
  - "Prof. Dr. Ion Chiricuta" Oncology Institute, Cluj-Napoca
  - S.C. Medisprof S.R.L., Cluj-Napoca
  - "Sfantul Nectarie" Oncology Center, Craiova
  - Oncomed SRL, Timișoara
- Russia (15):
  - RBHI "Kursk Regional Clinical Oncology Dispensary" of HCKR (legal address), Kursk, Kursk Oblast
  - RBHI "Kursk Regional Clinical Oncology Dispensary" of HCKR, Kursk, Kursk Oblast
  - Russian Research Center for Radiology and Surgical Technologies, Saint Petersburg, Pesochny
  - FSBI "Research Institute of Oncology n.a. N.N. Petrov" MoH RF, Saint Petersburg, Poselok Pesochniy
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - Scientific Research Institute of Urology named after N.A.Lopatkin of the Hersten Federal, Moscow
  - Moscow Scientific Research Oncology Institute n.a. P.A. Hertzen, Moscow
  - FBIH "Privolzhskiy Regional Medical Center" of FMBA, Nizhny Novgorod
  - SBIH of Nizhegorodskaya region "Clinical-Diagnostics center", Nizhny Novgorod
  - SBIH of Nizhegorodskaya region "Nizhniy Novgorod Regional Clinical Oncology Dispensary", Nizhny Novgorod
  - Clinical Hospital #122 n.a. L. G. Sokolov, Saint Petersburg
  - NS HI "Road Clinical Hospital of JSC "Russian Railways"", Saint Petersburg
  - LLC "Diagnostic center "Energo", Saint Petersburg
  - LLC "Clinical Diagnostic Center "Medex-pert", Yaroslavl
  - SHI YR Regional Clinical Oncology Hospital, Yaroslavl
- South Korea (15):
  - Clinical Trial Pharmacy, National Cancer Center, Goyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Clinical Pharmacy, Seongnam-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Kyungpook National University Medical Center, Clinical Pharmacy, Daegu
  - Kyungpook National University Medical Center, Daegu
  - Chungnam National University Hospital, Clinical Pharmacy, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Clinical Pharmacy, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Clinical Trial Pharmacy, Seoul
  - Samsung Medical Center Clinical Trial Pharmacy, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Sahlgrenska University Hospital, Dept of Oncology, Gothenburg, Sweden
- United Kingdom (14):
  - Cambridge University Hospital NHS Foundation Trust, Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Mount Vernon Cancer Centre, East & North Herts NHS Trust, London, Middlesex
  - Mount Vernon Cancer Centre, Pharmacy, London, Middlesex
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey, London
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Addenbrooke's Hospital, Central Pharmacy, Level 1, Cambridge
  - Beatson WOSCC, Glasgow
  - Beatson West of Scotland Cancer Centre, Gartnavel General Hospital,, Glasgow
  - St Bartholomew's Hospital, Barts Health NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Clinical Trials Pharmacy, The Christie, Manchester
  - Department of Medical Oncology, The Christie NHS Foundation Trust, Manchester
  - Academic Unit of Oncology, Nottingham University Hospitals NHS Trust-City Campus, Nottingham
  - Nottingham University Hospitals, Nottingham City Hospital, Nottingham Trials Pharmacy, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Tucker M, Chen YW, Voss MH, McGregor BA, Bilen MA, Grimm MO, Nathan P, Kollmannsberger C, Tomita Y, Huang B, Amezquita R, Mariani M, di Pietro A, Rini B. Association between neutrophil-to-eosinophil ratio and efficacy outcomes with avelumab plus axitinib or sunitinib in patients with advanced renal cell carcinoma: post hoc analyses from the JAVELIN Renal 101 trial. BMJ Oncol. 2024 Jun 12;3(1):e000181. doi: 10.1136/bmjonc-2023-000181. eCollection 2024. PMID 39886142
- [Derived] Grimm MO, Oya M, Choueiri TK, Motzer RJ, Schmidinger M, Quinn DI, Gravis-Mescam G, Verzoni E, Van den Eertwegh AJM, di Pietro A, Mariani M, Wang J, Thomaidou D, Albiges L. Impact of Prior Cytoreductive Nephrectomy on Efficacy in Patients with Synchronous Metastatic Renal Cell Carcinoma Treated with Avelumab plus Axitinib or Sunitinib: Post Hoc Analysis from the JAVELIN Renal 101 Phase 3 Trial. Eur Urol. 2024 Jan;85(1):8-12. doi: 10.1016/j.eururo.2023.09.016. Epub 2023 Oct 16. PMID 37852850
- [Derived] Rini BI, Atkins MB, Choueiri TK, Teresi RE, Rosbrook B, Thakur M, Hutson TE. Plain language summary looking at how long side effects last after treatment with axitinib is stopped in people with advanced renal cell carcinoma. Future Oncol. 2023 Dec;19(40):2623-2629. doi: 10.2217/fon-2023-0233. Epub 2023 Aug 1. PMID 37526095
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Haanen JBAG, Larkin J, Choueiri TK, Albiges L, Rini BI, Atkins MB, Schmidinger M, Penkov K, Michelon E, Wang J, Mariani M, di Pietro A, Motzer RJ. Extended follow-up from JAVELIN Renal 101: subgroup analysis of avelumab plus axitinib versus sunitinib by the International Metastatic Renal Cell Carcinoma Database Consortium risk group in patients with advanced renal cell carcinoma. ESMO Open. 2023 Jun;8(3):101210. doi: 10.1016/j.esmoop.2023.101210. Epub 2023 Apr 25. PMID 37104931
- [Derived] Rini BI, Moslehi JJ, Bonaca M, Schmidinger M, Albiges L, Choueiri TK, Motzer RJ, Atkins MB, Haanen J, Mariani M, Wang J, Hariharan S, Larkin J. Prospective Cardiovascular Surveillance of Immune Checkpoint Inhibitor-Based Combination Therapy in Patients With Advanced Renal Cell Cancer: Data From the Phase III JAVELIN Renal 101 Trial. J Clin Oncol. 2022 Jun 10;40(17):1929-1938. doi: 10.1200/JCO.21.01806. Epub 2022 Mar 3. PMID 35239416
- [Derived] Masters JC, Khandelwal A, di Pietro A, Dai H, Brar S. Model-informed drug development supporting the approval of the avelumab flat-dose regimen in patients with advanced renal cell carcinoma. CPT Pharmacometrics Syst Pharmacol. 2022 Apr;11(4):458-468. doi: 10.1002/psp4.12771. Epub 2022 Feb 27. PMID 35166465
- [Derived] Rini BI, Atkins MB, Choueiri TK, Thomaidou D, Rosbrook B, Thakur M, Hutson TE. Time to Resolution of Axitinib-Related Adverse Events After Treatment Interruption in Patients With Advanced Renal Cell Carcinoma. Clin Genitourin Cancer. 2021 Oct;19(5):e306-e312. doi: 10.1016/j.clgc.2021.03.019. Epub 2021 Apr 5. PMID 33947608
- [Derived] Choueiri TK, Larkin J, Pal S, Motzer RJ, Rini BI, Venugopal B, Alekseev B, Miyake H, Gravis G, Bilen MA, Hariharan S, Chudnovsky A, Ching KA, Mu XJ, Mariani M, Robbins PB, Huang B, di Pietro A, Albiges L. Efficacy and correlative analyses of avelumab plus axitinib versus sunitinib in sarcomatoid renal cell carcinoma: post hoc analysis of a randomized clinical trial. ESMO Open. 2021 Jun;6(3):100101. doi: 10.1016/j.esmoop.2021.100101. Epub 2021 Apr 23. PMID 33901870
- [Derived] Motzer RJ, Robbins PB, Powles T, Albiges L, Haanen JB, Larkin J, Mu XJ, Ching KA, Uemura M, Pal SK, Alekseev B, Gravis G, Campbell MT, Penkov K, Lee JL, Hariharan S, Wang X, Zhang W, Wang J, Chudnovsky A, di Pietro A, Donahue AC, Choueiri TK. Avelumab plus axitinib versus sunitinib in advanced renal cell carcinoma: biomarker analysis of the phase 3 JAVELIN Renal 101 trial. Nat Med. 2020 Nov;26(11):1733-1741. doi: 10.1038/s41591-020-1044-8. Epub 2020 Sep 7. PMID 32895571
- [Derived] Choueiri TK, Motzer RJ, Rini BI, Haanen J, Campbell MT, Venugopal B, Kollmannsberger C, Gravis-Mescam G, Uemura M, Lee JL, Grimm MO, Gurney H, Schmidinger M, Larkin J, Atkins MB, Pal SK, Wang J, Mariani M, Krishnaswami S, Cislo P, Chudnovsky A, Fowst C, Huang B, di Pietro A, Albiges L. Updated efficacy results from the JAVELIN Renal 101 trial: first-line avelumab plus axitinib versus sunitinib in patients with advanced renal cell carcinoma. Ann Oncol. 2020 Aug;31(8):1030-1039. doi: 10.1016/j.annonc.2020.04.010. Epub 2020 Apr 25. PMID 32339648
- [Derived] Motzer RJ, Penkov K, Haanen J, Rini B, Albiges L, Campbell MT, Venugopal B, Kollmannsberger C, Negrier S, Uemura M, Lee JL, Vasiliev A, Miller WH Jr, Gurney H, Schmidinger M, Larkin J, Atkins MB, Bedke J, Alekseev B, Wang J, Mariani M, Robbins PB, Chudnovsky A, Fowst C, Hariharan S, Huang B, di Pietro A, Choueiri TK. Avelumab plus Axitinib versus Sunitinib for Advanced Renal-Cell Carcinoma. N Engl J Med. 2019 Mar 21;380(12):1103-1115. doi: 10.1056/NEJMoa1816047. Epub 2019 Feb 16. PMID 30779531
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 886 participants were enrolled and randomized in the study.
Groups:
- Avelumab + Axitinib: Participants with advanced renal cell carcinoma (aRCC) received avelumab 10 milligram per kilogram (mg/kg), intravenously (IV) once every two weeks (Q2W) in a 6-week cycle plus axitinib 5 mg, orally twice daily (BID). Each treatment cycle was of 42 days.
- Sunitinib: Participants with aRCC received sunitinib 50 mg orally, QD on a schedule of 4 weeks on treatment followed by 2 weeks off treatment (schedule 4/2 in 6-week cycles). Each treatment cycle was of 42 days.
Period: Overall Study
Arm/Group | Avelumab + Axitinib | Sunitinib
Started | 442 | 444
Completed | 0 | 0
Not Completed | 442 | 444
Not completed — Other | 18 | 6
Not completed — Protocol Violation | 2 | 1
Not completed — Non-compliance with study drug | 1 | 1
Not completed — No longer met eligibility criteria | 6 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 25 | 22
Not completed — Global deterioration of health status | 18 | 20
Not completed — Physician Decision | 15 | 8
Not completed — Adverse Event | 86 | 65
Not completed — Withdrawal by Subject | 29 | 43
Not completed — Progressive disease | 236 | 266
Not completed — Participation terminated by sponsor | 6 | 9

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Avelumab + Axitinib: Participants with aRCC received avelumab 10 mg/kg, IV at Q2W in a 6-week cycle plus axitinib 5 mg, orally BID. Each treatment cycle was of 42 days.
- Total: Total of all reporting groups
Arm/Group | Avelumab + Axitinib | Sunitinib | Total
Number analyzed (Participants) | 442 | 444 | 886
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.86 (9.95) | 60.66 (10.28) | 60.76 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 100 | 226
  Male | 316 | 344 | 660
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 37
  Not Hispanic or Latino | 388 | 377 | 765
  Unknown or Not Reported | 35 | 49 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 70 | 63 | 133
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 10 | 20
  White | 332 | 334 | 666
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 26 | 32 | 58

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) in Programmed Death-Ligand 1 (PD-L1) Positive Participants
Description: PFS: time from the date of randomization to the date of the first documentation of progressive disease (PD) according to Response Evaluation Criteria in Solid Tumours (RECIST version [v] 1.1) or death due to any cause, whichever occurred first as assessed by BICR. PFS data was censored on date of last adequate tumor assessment for participants who did not have an event (PD or death), who started new anti-cancer therapy prior to an event or for participants with an event after 2 or more missing tumor assessments.
  PD was defined as at least a 20 percent (%), increase in the sum of all the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to relative increase of 20 %, sum must have also demonstrated an absolute more than (>) of at least 5 millimeter (mm). The appearance of one or more new lesions was also considered progression.
Time Frame: From date of randomization to the first documentation of PD or death due to any cause or censoring date, whichever occurred first (maximum up to approximately 26 months)
Population: FAS included all participants who were randomized. Analysis was performed on subset of randomized participants, who were PD-L1 positive.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Avelumab + Axitinib: Participants with aRCC received avelumab 10 mg/kg, IV at Q2W in a 6-week cycle plus axitinib 5 mg, orally BID. Each treatment cycle was 42 days.
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 270 | 290
Months | 13.8 [11.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with event. | 7.2 [5.7 to 9.7]
Statistical Analysis 1: Comparison: Avelumab + Axitinib vs Sunitinib; Test type: Superiority; p = 0.0001, Log Rank — 2-sided p-value; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.475 to 0.790]

2. Primary Outcome: Overall Survival (OS) in PD-L1 Positive Participants
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From the date of randomization to the date of death due to any cause or censoring date, whichever occurred first (maximum up to approximately 89 months)
Population: FAS included all participants who are randomized. Analysis was performed on subset of randomized participants, who were PD-L1 positive.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 270 | 290
Months | 43.2 [36.5 to 51.7] | 36.2 [29.8 to 44.2]
Statistical Analysis 1: Comparison: Avelumab + Axitinib vs Sunitinib; Test type: Superiority; p = 0.1509, Log Rank — 2-sided p-value; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.701 to 1.057]

3. Secondary Outcome: PFS as Assessed by BICR in Participants Irrespective of PD-L1 Expression
Description: PFS: time from the date of randomization to the date of the first documentation of PD or death due to any cause, whichever occurred first as assessed by BICR. PFS data was censored on date of last adequate tumor assessment for participants who did not have an event (PD or death), who started new anti-cancer therapy prior to an event or for participants with an event after 2 or more missing tumor assessments. PD was defined as at least a 20% increase in the sum of all the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to relative increase of 20 %, sum must have also demonstrated an absolute > of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: as for outcome 1
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Months | 13.8 [11.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with event. | 8.4 [6.9 to 11.1]
Statistical Analysis 1: Comparison: Avelumab + Axitinib vs Sunitinib; Test type: Superiority; p = 0.0002, Log Rank — 2-sided p-value; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.563 to 0.840]

4. Secondary Outcome: OS in Participants Irrespective of PD-L1 Expression
Description: OS was defined as the time (in months) from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: as for outcome 2
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Months | 44.8 [39.7 to 51.1] | 38.9 [31.4 to 45.2]
Statistical Analysis 1: Comparison: Avelumab + Axitinib vs Sunitinib; Test type: Superiority; p = 0.1338, Log Rank — 2-sided p-value; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.749 to 1.039]

5. Secondary Outcome: Percentage of Participants With Objective Response (OR) as Assessed by BICR Irrespective of PD-L1 Expression
Description: OR was defined as best overall response of complete response (CR) or partial response (PR) according to RECIST v1.1 as assessed by BICR recorded from date of randomization until disease progression. CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed. 95% CI was based on Clopper-Pearson method.
Time Frame: From date of randomization until PD (maximum up to approximately 26 months)
Population: FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Percentage of participants | 51.4 [46.6 to 56.1] | 25.7 [21.7 to 30.0]

6. Secondary Outcome: Percentage of Participants With OR as Assessed by Investigator Irrespective of PD-L1 Expression
Description: OR was defined as best overall response of CR or PR according to RECIST v1.1 as assessed by investigator recorded from date of randomization until disease progression. CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed. 95% CI was based on Clopper-Pearson method.
Time Frame: From date of randomization until PD (maximum up to approximately 89 months)
Population: FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Percentage of participants | 59.7 [55.0 to 64.3] | 32.0 [27.7 to 36.5]

7. Secondary Outcome: Percentage of Participants With Disease Control (DC) as Assessed by BICR Irrespective of PD-L1 Expression
Description: DC was defined as a best overall response of CR, PR, non-CR/non-PD or stable disease (SD) according to RECIST v1.1 as assessed by BICR. CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. All lymph nodes must decrease to normal size (short axis<10mm). PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. Non-CR/Non-PD was defined as persistence of any non-target lesions and/or tumor marker level above the normal limits. SD was defined as not to qualify for CR, PR or PD for target lesions and followed PR only if the sum increased by less than 20% from the nadir (smallest sum of diameters consider baseline and all assessments prior to the time point under evaluation), but enough that a previously documented 30% decrease no longer holds.
Time Frame: From date of randomization until PD (maximum up to approximately 26 months)
Population: FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Percentage of participants | 82.8 [79.0 to 86.2] | 73.4 [69.1 to 77.5]

8. Secondary Outcome: Percentage of Participants With DC as Assessed by Investigator Irrespective of PD-L1 Expression
Description: DC was defined as a best overall response of CR, PR, non-CR/non-PD or SD according to RECIST v1.1 as assessed by investigator. CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. All lymph nodes must decrease to normal size (short axis<10mm). PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. Non-CR/Non-PD was defined as persistence of any non-target lesions and/or tumor marker level above the normal limits. SD was defined as not to qualify for CR, PR or PD for target lesions and followed PR only if the sum increased by less than 20% from the nadir (smallest sum of diameters consider baseline and all assessments prior to the time point under evaluation), but enough that a previously documented 30% decrease no longer holds.
Time Frame: From date of randomization until PD (maximum up to approximately 89 months)
Population: FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Percentage of participants | 85.1 [81.4 to 88.3] | 76.4 [72.1 to 80.2]

9. Secondary Outcome: Time to Tumor Response (TTR) as Assessed by BICR in Participants Irrespective of PD-L1 Expression
Description: TTR was defined as the time from randomization to the first documentation of objective tumor response according to RECIST v1.1 as assessed by BICR (CR or PR) which is subsequently confirmed. CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed.
Time Frame: From the date of randomization to the first documentation of objective response (CR or PR) (maximum up to approximately 26 months)
Population: FAS included all randomized participants. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 227 | 114
Months | 2.6 [1.2 to 13.8] | 3.2 [1.2 to 11.6]

10. Secondary Outcome: TTR as Assessed by Investigator in Participants Irrespective of PD-L1 Expression
Description: TTR was defined as the time from randomization to the first documentation of objective tumor response according to RECIST v1.1 as assessed by investigator (CR or PR) which is subsequently confirmed. CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed.
Time Frame: From the date of randomization to the first documentation of objective response (CR or PR) (maximum up to approximately 89 months)
Population: as for outcome 9
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 264 | 142
Months | 2.8 [1.1 to 34.5] | 2.8 [1.2 to 65.2]

11. Secondary Outcome: Duration of Response (DR) as Assessed by BICR in Participants Irrespective of PD-L1 Expression
Description: BICR assessed DR: time from first documentation of OR (confirmed CR or PR) to date of first documentation of objective tumor progression assessed by BICR or death due to any cause whichever occurred first. As per RECIST v1.1. CR: complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed. PD: at least a 20% increase in the sum of all the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to relative increase of 20%, sum must have also demonstrated an absolute > of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From documentation of OR until date of first documentation of PD or death due to any cause, whichever occurred first (maximum up to approximately 26 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 227 | 114
Months | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of participants with event. | NA [11.2 to NA] — Median and upper limit of 95% CI was not estimable due to insufficient number of participants with event.

12. Secondary Outcome: DR as Assessed by Investigator in Participants Irrespective of PD-L1 Expression
Description: Investigator assessed DR: time from first documentation of OR (confirmed CR or PR) to date of first documentation of objective tumor progression (PD) assessed by investigator or death due to any cause whichever occurred first. As per RECIST v1.1. CR: complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed. PD: at least a 20% increase in the sum of all the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to relative increase of 20%, sum must have also demonstrated an absolute > of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From documentation of OR until date of first documentation of PD or death due to any cause, whichever occurred first (maximum up to approximately 89 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 264 | 142
Months | 19.4 [16.4 to 22.3] | 14.5 [8.7 to 16.6]

13. Secondary Outcome: PFS as Assessed by Investigator in Participants Irrespective of PD-L1 Expression
Description: Investigator assessed PFS: time from the date of randomization to the date of the first documentation of PD according to RECIST v1.1 or death due to any cause, whichever occurred first. PFS data was censored on date of last adequate tumor assessment for participants who did not have an event (PD or death), who started new anti-cancer therapy prior to an event or for participants with an event after 2 or more missing tumor assessments. PD was defined as at least a 20% increase in the sum of all the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to relative increase of 20 %, sum must have also demonstrated an absolute > of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From date of randomization until PD, whichever occurred first (maximum up to approximately 89 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Months | 13.9 [11.1 to 16.6] | 8.5 [8.2 to 9.7]
Statistical Analysis 1: Comparison: Avelumab + Axitinib vs Sunitinib; Test type: Superiority; p < .0001, Log Rank — 2-sided p-value; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.565 to 0.768]

14. Secondary Outcome: Progression-Free Survival on Next-line Therapy (PFS2) in Participants Irrespective of PD-L1 Expression
Description: PFS2 is defined as the time (in months) from randomization to discontinuation of next-line treatment after first objective disease progression by investigator assessment, second objective disease progression by investigator assessment after initiation of next-line treatment, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the sum of all the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to relative increase of 20 %, sum must have also demonstrated an absolute > of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From date of randomization until PD or death, whichever occurred first (maximum up to approximately 89 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Months | 30.4 [25.8 to 34.6] | 19.4 [17.0 to 22.4]
Statistical Analysis 1: Comparison: Avelumab + Axitinib vs Sunitinib; Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.551 to 0.754]

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) Graded Based on National Cancer Institute -Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version (V) 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were those events with onset dates occurring during the on-treatment period for the first time, or if the worsening of an event was during the on-treatment period (time from the first dose of study treatment through 90 days after last dose of study treatment or start day of new anti-cancer drug therapy-1 day). As per NCI-CTCAE v4.03, grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death.
Time Frame: From start of study treatment until 90 days after last dose of study treatment (maximum up to approximately 92 months)
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 434 | 439
Participants
  Grade 1 | 5 | 17
  Grade 2 | 64 | 73
  Grade 3 | 271 | 268
  Grade 4 | 64 | 54
  Grade 5 | 30 | 24

16. Secondary Outcome: Number of Participants According to Grade Shift in Hematology Parameters
Description: Following hematology parameters were assessed: hemoglobin decreased (anemia), hemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased and white blood cell (WBC) decreased. Laboratory abnormalities were graded as per NCI- CTCAE v 4.03 where, grade(G) 0= non-missing lab value that does not meet either of G1 through 4 criteria, G1=mild, G2=moderate, G3=severe, G4=life-threatening consequences and G5=death. Baseline was defined as last assessment prior to first dose of study treatment. Number of participants with a baseline grade of 0 to 4 which shifted to G3-4 post-baseline are reported in this outcome measure. Only non-zero categories for any reporting arm are reported.
Time Frame: From start of study treatment until 90 days after last dose of study treatment (maximum up to approximately 92 months)
Population: Safety analysis set included all participants who received at least one dose of study drug. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 428 | 434
Participants
  Anemia (Baseline G0 to post-baseline G3-4) | 3 | 9
  Anemia (Baseline G1 to post-baseline G3-4) | 6 | 21
  Anemia (Baseline G2 to post-baseline G3-4) | 4 | 14
  Anemia (Baseline G3 to post-baseline G3-4) | 0 | 2
  Lymphocytes count decreased (Baseline G0 to post-baseline G3-4) | 21 | 53
  Lymphocytes count decreased (Baseline G1 to post-baseline G3-4) | 11 | 18
  Lymphocytes count decreased (Baseline G2 to post-baseline G3-4) | 7 | 15
  Lymphocytes count decreased (Baseline G3 to post-baseline G3-4) | 2 | 6
  Neutrophils count decreased (Baseline G0 to post-baseline G3-4) | 7 | 108
  Neutrophils count decreased (Baseline G1 to post-baseline G3-4) | 0 | 2
  Neutrophils count decreased (Baseline G2 to post-baseline G3-4) | 0 | 1
  Platelets count decreased (Baseline G0 to post-baseline G3-4) | 3 | 61
  Platelets count decreased (Baseline G1 to post-baseline G3-4) | 1 | 6
  WBC decreased (Baseline G0 to post-baseline G3-4) | 1 | 35
  WBC decreased (Baseline G1 to post-baseline G3-4) | 0 | 7
  WBC decreased (Baseline G2 to post-baseline G3-4) | 0 | 2

17. Secondary Outcome: Number of Participants According to Grade Shift in Chemistry Parameters
Description: Following chemistry parameters were assessed: alanine aminotransferase(ALT) increased, alkaline phosphatase(ALP) increased, aspartate aminotransferase(AST) increased, blood bilirubin increased, cholesterol high, creatinine phosphokinase(CPK) increased, creatinine increased, gamma glutamyl transferase(GGT) increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesmia, hypernatremia, hypertriglyceridemia, hypoalbuminemia, hypokalemia, hypomagnesemia, hyponatremia, lipase increased and serum amylase increased. Laboratory abnormality graded as per NCI CTCAE v4.03; G0=non-missing lab value that does not meet either of G1 through 4 criteria, G1=mild, G2=moderate, G3=severe, G4=life-threatening consequences and G5=death. Number of participants with a baseline grade of 0 to 4 which shifted to G3-4 post-baseline are reported. Only non-zero categories for any reporting arm are reported.
Time Frame: From start of study treatment until 90 days after last dose of study treatment (maximum up to approximately 92 months)
Population: Safety analysis set included all participants who received at least one dose of study drug. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. "Number Analyzed" signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 428 | 433
Participants
  ALT increased (Baseline G0 to post-baseline G3-4) | 42 | 19
  ALT increased (Baseline G1 to post-baseline G3-4) | 3 | 0
  ALP increased (Baseline G0 to post-baseline G3-4) | 9 | 0
  ALP increased (Baseline G1 to post-baseline G3-4) | 5 | 6
  ALP increased (Baseline G2 to post-baseline G3-4) | 1 | 3
  ALP increased (Baseline G3 to post-baseline G3-4) | 4 | 1
  AST increased (Baseline G0 to post-baseline G3-4) | 26 | 16
  AST increased (Baseline G1 to post-baseline G3-4) | 6 | 4
  AST increased (Baseline G3 to post-baseline G3-4) | 1 | 0
  Blood bilirubin increased (Baseline G0 to post-baseline G3-4) | 3 | 6
  Blood bilirubin increased (Baseline G1 to post-baseline G3-4) | 2 | 0
  Cholesterol high (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 419 | 413
  Cholesterol high (Baseline G0 to post-baseline G3-4) | 8 | 3
  Cholesterol high (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 419 | 413
  Cholesterol high (Baseline G1 to post-baseline G3-4) | 4 | 3
  Cholesterol high (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 419 | 413
  Cholesterol high (Baseline G2 to post-baseline G3-4) | 0 | 1
  CPK increased (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 417 | 415
  CPK increased (Baseline G0 to post-baseline G3-4) | 7 | 7
  CPK increased (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 417 | 415
  CPK increased (Baseline G2 to post-baseline G3-4) | 0 | 1
  CPK increased (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 417 | 415
  CPK increased (Baseline G1 to post-baseline G3-4) | 0 | 2
  CPK increased (Baseline G3 to post-baseline G3-4): number analyzed (Participants) | 417 | 415
  CPK increased (Baseline G3 to post-baseline G3-4) | 1 | 0
  Creatinine increased (Baseline G0 to post-baseline G3-4) | 7 | 2
  Creatinine increased (Baseline G1 to post-baseline G3-4) | 4 | 5
  Creatinine increased (Baseline G2 to post-baseline G3-4) | 0 | 1
  Creatinine increased (Baseline G3 to post-baseline G3-4) | 0 | 1
  GGT increased (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 419 | 415
  GGT increased (Baseline G0 to post-baseline G3-4) | 15 | 16
  GGT increased (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 419 | 415
  GGT increased (Baseline G1 to post-baseline G3-4) | 20 | 7
  GGT increased (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 419 | 415
  GGT increased (Baseline G2 to post-baseline G3-4) | 12 | 4
  GGT increased (Baseline G3 to post-baseline G3-4): number analyzed (Participants) | 419 | 415
  GGT increased (Baseline G3 to post-baseline G3-4) | 7 | 2
  GGT increased (Baseline G4 to post-baseline G3-4): number analyzed (Participants) | 419 | 415
  GGT increased (Baseline G4 to post-baseline G3-4) | 0 | 1
  Hypercalcemia (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypercalcemia (Baseline G0 to post-baseline G3-4) | 4 | 4
  Hypercalcemia (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypercalcemia (Baseline G1 to post-baseline G3-4) | 1 | 2
  Hypercalcemia (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypercalcemia (Baseline G2 to post-baseline G3-4) | 1 | 1
  Hypercalcemia (Baseline G3 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypercalcemia (Baseline G3 to post-baseline G3-4) | 0 | 2
  Hypercalcemia (Baseline G4 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypercalcemia (Baseline G4 to post-baseline G3-4) | 0 | 1
  Hyperglycemia (Baseline G0 to post-baseline G3-4) | 37 | 20
  Hyperglycemia (Baseline G1 to post-baseline G3-4) | 4 | 3
  Hyperglycemia (Baseline G2 to post-baseline G3-4) | 5 | 3
  Hyperglycemia (Baseline G3 to post-baseline G3-4) | 6 | 4
  Hyperkalemia (Baseline G0 to post-baseline G3-4) | 19 | 16
  Hyperkalemia (Baseline G1 to post-baseline G3-4) | 1 | 5
  Hyperkalemia (Baseline G2 to post-baseline G3-4) | 3 | 3
  Hyperkalemia (Baseline G3 to post-baseline G3-4) | 1 | 0
  Hyperkalemia (Baseline G4 to post-baseline G3-4) | 0 | 1
  Hypermagnesemia (Baseline G0 to post-baseline G3-4) | 13 | 20
  Hypermagnesemia (Baseline G1 to post-baseline G3-4) | 1 | 2
  Hypernatremia (Baseline G0 to post-baseline G3-4) | 7 | 2
  Hypertriglyceridemia (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 419 | 411
  Hypertriglyceridemia (Baseline G0 to post-baseline G3-4) | 18 | 3
  Hypertriglyceridemia (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 419 | 411
  Hypertriglyceridemia (Baseline G1 to post-baseline G3-4) | 31 | 23
  Hypertriglyceridemia (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 419 | 411
  Hypertriglyceridemia (Baseline G2 to post-baseline G3-4) | 15 | 6
  Hypertriglyceridemia (Baseline G3 to post-baseline G3-4): number analyzed (Participants) | 419 | 411
  Hypertriglyceridemia (Baseline G3 to post-baseline G3-4) | 4 | 5
  Hypertriglyceridemia (Baseline G4 to post-baseline G3-4): number analyzed (Participants) | 419 | 411
  Hypertriglyceridemia (Baseline G4 to post-baseline G3-4) | 0 | 1
  Hypoalbunemia (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypoalbunemia (Baseline G0 to post-baseline G3-4) | 3 | 6
  Hypoalbunemia (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypoalbunemia (Baseline G1 to post-baseline G3-4) | 1 | 1
  Hypoalbunemia (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypoalbunemia (Baseline G2 to post-baseline G3-4) | 2 | 2
  Hypoalbunemia (Baseline G3 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypoalbunemia (Baseline G3 to post-baseline G3-4) | 1 | 2
  Hypocalcemia (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypocalcemia (Baseline G0 to post-baseline G3-4) | 4 | 4
  Hypocalcemia (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypocalcemia (Baseline G1 to post-baseline G3-4) | 0 | 1
  Hypocalcemia (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 418 | 419
  Hypocalcemia (Baseline G2 to post-baseline G3-4) | 1 | 0
  Hypoglycemia (Baseline G0 to post-baseline G3-4) | 2 | 1
  Hypokalemia (Baseline G0 to post-baseline G3-4) | 17 | 15
  Hypokalemia (Baseline G2 to post-baseline G3-4) | 2 | 1
  Hypomagnesemia (Baseline G0 to post-baseline G3-4) | 3 | 1
  Hypomagnesemia (Baseline G1 to post-baseline G3-4) | 2 | 1
  Hypomagnesemia (Baseline G2 to post-baseline G3-4) | 1 | 0
  Hyponatremia (Baseline G0 to post-baseline G3-4) | 42 | 35
  Hyponatremia (Baseline G1 to post-baseline G3-4) | 19 | 14
  Hyponatremia (Baseline G3 to post-baseline G3-4) | 1 | 2
  Lipase increased (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 419 | 414
  Lipase increased (Baseline G0 to post-baseline G3-4) | 63 | 27
  Lipase increased (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 419 | 414
  Lipase increased (Baseline G1 to post-baseline G3-4) | 19 | 8
  Lipase increased (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 419 | 414
  Lipase increased (Baseline G2 to post-baseline G3-4) | 7 | 3
  Lipase increased (Baseline G3 to post-baseline G3-4): number analyzed (Participants) | 419 | 414
  Lipase increased (Baseline G3 to post-baseline G3-4) | 2 | 7
  Lipase increased (Baseline G4 to post-baseline G3-4): number analyzed (Participants) | 419 | 414
  Lipase increased (Baseline G4 to post-baseline G3-4) | 1 | 0
  Serum amylase increased (Baseline G0 to post-baseline G3-4): number analyzed (Participants) | 412 | 407
  Serum amylase increased (Baseline G0 to post-baseline G3-4) | 21 | 4
  Serum amylase increased (Baseline G1 to post-baseline G3-4): number analyzed (Participants) | 412 | 407
  Serum amylase increased (Baseline G1 to post-baseline G3-4) | 12 | 4
  Serum amylase increased (Baseline G2 to post-baseline G3-4): number analyzed (Participants) | 412 | 407
  Serum amylase increased (Baseline G2 to post-baseline G3-4) | 4 | 4
  Serum amylase increased (Baseline G3 to post-baseline G3-4): number analyzed (Participants) | 412 | 407
  Serum amylase increased (Baseline G3 to post-baseline G3-4) | 1 | 3

18. Secondary Outcome: Change From Baseline in Vital Signs - Blood Pressure at Day 1 of Cycle 2, 3, 4, 5, 6, 7 and End of Treatment (EOT) Visit
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured with the participant in the seated position after the participant had been sitting quietly for at least 5 minutes.
Time Frame: Baseline (pre-dose on Day 1 of Cycle 1), Day 1 of Cycle 2, 3, 4, 5, 6, 7, EOT visit (maximum up to approximately 89 months) (each cycle=42 days)
Population: Safety analysis set included all participants who received at least one dose of study drug. "Number Analyzed" signifies number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 434 | 439
Millimeters of mercury
  Baseline: Sitting SBP | 126.5 (13.52) | 126.3 (12.00)
  Change at Cycle 2, Day 1: Sitting SBP: number analyzed (Participants) | 380 | 344
  Change at Cycle 2, Day 1: Sitting SBP | 4.7 (16.08) | 0.8 (12.49)
  Change at Cycle 3, Day 1: Sitting SBP: number analyzed (Participants) | 363 | 310
  Change at Cycle 3, Day 1: Sitting SBP | 3.8 (16.43) | 1.2 (12.81)
  Change at Cycle 4, Day 1: Sitting SBP: number analyzed (Participants) | 342 | 271
  Change at Cycle 4, Day 1: Sitting SBP | 3.0 (15.95) | 0.1 (13.01)
  Change at Cycle 5, Day 1: Sitting SBP: number analyzed (Participants) | 332 | 244
  Change at Cycle 5, Day 1: Sitting SBP | 2.5 (15.42) | -0.1 (12.26)
  Change at Cycle 6, Day 1: Sitting SBP: number analyzed (Participants) | 310 | 215
  Change at Cycle 6, Day 1: Sitting SBP | 1.6 (15.39) | -0.1 (12.97)
  Change at Cycle 7, Day 1: Sitting SBP: number analyzed (Participants) | 282 | 191
  Change at Cycle 7, Day 1: Sitting SBP | 1.9 (15.39) | 0.4 (13.56)
  Change at End of Treatment: Sitting SBP: number analyzed (Participants) | 205 | 273
  Change at End of Treatment: Sitting SBP | 0.9 (17.40) | 1.7 (15.67)
  Baseline: Sitting DBP | 75.7 (9.32) | 75.9 (9.41)
  Change at Cycle 2, Day 1: Sitting DBP: number analyzed (Participants) | 380 | 344
  Change at Cycle 2, Day 1: Sitting DBP | 5.8 (10.92) | -0.1 (8.60)
  Change at Cycle 3, Day 1: Sitting DBP: number analyzed (Participants) | 363 | 310
  Change at Cycle 3, Day 1: Sitting DBP | 4.9 (10.98) | 0.0 (9.64)
  Change at Cycle 4, Day 1: Sitting DBP: number analyzed (Participants) | 342 | 271
  Change at Cycle 4, Day 1: Sitting DBP | 4.8 (11.61) | -1.9 (9.30)
  Change at Cycle 5, Day 1: Sitting DBP: number analyzed (Participants) | 332 | 244
  Change at Cycle 5, Day 1: Sitting DBP | 4.5 (11.17) | -1.9 (9.71)
  Change at Cycle 6, Day 1: Sitting DBP: number analyzed (Participants) | 310 | 215
  Change at Cycle 6, Day 1: Sitting DBP | 3.8 (10.18) | -1.3 (9.89)
  Change at Cycle 7, Day 1: Sitting DBP: number analyzed (Participants) | 282 | 191
  Change at Cycle 7, Day 1: Sitting DBP | 3.8 (11.04) | -1.1 (9.90)
  Change at End of Treatment: Sitting DBP: number analyzed (Participants) | 205 | 273
  Change at End of Treatment: Sitting DBP | 1.5 (12.70) | -0.9 (10.92)

19. Secondary Outcome: Change From Baseline in Vital Signs - Pulse Rate at Day 1 of Cycle 2, 3, 4, 5, 6, 7 and EOT Visit
Description: Pulse rate was measured with the participant in the seated position after the participant had been sitting quietly for at least 5 minutes.
Time Frame: as for outcome 18
Population: Safety analysis set included all participants who received at least one dose of study drug. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. "Number Analyzed" signifies number of participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 433 | 439
beats per minute
  Baseline | 75.4 (12.49) | 75.6 (12.63)
  Change at Cycle 2, Day 1: number analyzed (Participants) | 347 | 319
  Change at Cycle 2, Day 1 | 0.4 (12.77) | 3.1 (10.69)
  Change at Cycle 3, Day 1: number analyzed (Participants) | 338 | 289
  Change at Cycle 3, Day 1 | 0.8 (12.58) | 3.1 (11.34)
  Change at Cycle 4, Day 1: number analyzed (Participants) | 327 | 244
  Change at Cycle 4, Day 1 | -0.6 (12.79) | 2.8 (10.34)
  Change at Cycle 5, Day 1: number analyzed (Participants) | 319 | 227
  Change at Cycle 5, Day 1 | -0.5 (12.00) | 2.5 (10.82)
  Change at Cycle 6, Day 1: number analyzed (Participants) | 299 | 203
  Change at Cycle 6, Day 1 | -1.9 (12.37) | 1.6 (10.75)
  Change at Cycle 7, Day 1: number analyzed (Participants) | 269 | 182
  Change at Cycle 7, Day 1 | -1.9 (11.69) | 2.1 (10.13)
  Change at End of Treatment: number analyzed (Participants) | 196 | 250
  Change at End of Treatment | 2.9 (15.29) | 3.5 (12.27)

20. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to Toxicity
Description: Number of participants who discontinued treatment due to toxicity are reported in this outcome measure.
Time Frame: From first dose of study treatment until discontinuation of study treatment (maximum up to approximately 89 months)
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 434 | 439
Participants | 136 [lower limit 17.41] | 65 [lower limit 12.82]

21. Secondary Outcome: Time to Treatment Discontinuation/Failure Due to Toxicity
Description: Time to treatment discontinuation/ failure due to toxicity was defined as the time from first dose of study treatment to discontinuation of study treatment due to an adverse event or death due to study treatment toxicity.
Time Frame: From first dose of study treatment until discontinuation of study treatment (maximum up to approximately 89 months)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 136 | 65
Months | 13.5 (17.41) | 10.5 (12.82)

22. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Avelumab
Description: Predose concentration during multiple dosing.
Time Frame: Pre dose (0 hour) on Day 1, 15 and 29 of Cycle 1, Day 1 and 29 of Cycles 2, 3, 4 and Day 1 of Cycle 6
Population: Avelumab PK concentration analysis set: all participants who had at least one post-dose concentration above lower limit of quantitation (LLQ) for avelumab. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. "Number Analyzed" signifies number of participants evaluable for the specified rows. This outcome measure was not planned to be analyzed in ''Sunitinib'' reporting group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 389
Micrograms per milliliter
  Cycle 1 (day 1) | 4.218 (1232)
  Cycle 1 (day 15): number analyzed (Participants) | 267
  Cycle 1 (day 15) | 18.69 (102)
  Cycle 1 (day 29): number analyzed (Participants) | 270
  Cycle 1 (day 29) | 21.99 (96)
  Cycle 2 (day 1): number analyzed (Participants) | 314
  Cycle 2 (day 1) | 24.87 (92)
  Cycle 2 (day 29): number analyzed (Participants) | 215
  Cycle 2 (day 29) | 22.62 (113)
  Cycle 3 (day 1): number analyzed (Participants) | 202
  Cycle 3 (day 1) | 26.04 (98)
  Cycle 3 (day 29): number analyzed (Participants) | 181
  Cycle 3 (day 29) | 30.13 (82)
  Cycle 4 (day 1): number analyzed (Participants) | 186
  Cycle 4 (day 1) | 29.15 (98)
  Cycle 4 (day 29): number analyzed (Participants) | 160
  Cycle 4 (day 29) | 31.38 (86)
  Cycle 6 (day 1): number analyzed (Participants) | 130
  Cycle 6 (day 1) | 39.11 (58)

23. Secondary Outcome: Ctrough of Axitinib
Description: Predose concentration during multiple dosing.
Time Frame: Pre dose (0 hour) on day 15 and 29 of cycle 1 (each cycle= 6 weeks)
Population: Axitinib PK concentration analysis set: all participants who received at least one dose of study drug and have at least one post-dose concentration above lower limit of quantitation (LLQ) for axitinib. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies number of participants evaluable for the specified rows. This outcome measure was not planned to be analyzed in ''Sunitinib'' reporting group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 312
Nanograms per milliliter
  Cycle1 (day 15) | 4.904 (172)
  Cycle1 (day 29): number analyzed (Participants) | 302
  Cycle1 (day 29) | 6.272 (174)

24. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Axitinib
Time Frame: 2 hours post-dose on Day 1, pre-dose and 2 hours post dose on Days 15 and 29 of Cycle 1
Population: Axitinib PK concentration analysis: all participants who received at least one dose of study drug and have at least one post-dose concentration above lower limit of quantitation (LLQ) for axitinib. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. "Number Analyzed" signifies number of participants evaluable for the specified rows. This outcome measure was not planned to be analyzed in ''Sunitinib'' reporting group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 316
Nanogram per milliliter
  Cycle1 (day 1); Post Dose | 17.93 (182)
  Cycle1 (day 15); Pre-Dose: number analyzed (Participants) | 312
  Cycle1 (day 15); Pre-Dose | 4.904 (172)
  Cycle1 (day 15); Post Dose: number analyzed (Participants) | 286
  Cycle1 (day 15); Post Dose | 18.45 (157)
  Cycle1 (day 29); Pre-Dose: number analyzed (Participants) | 302
  Cycle1 (day 29); Pre-Dose | 6.272 (174)
  Cycle1 (day 29); Post Dose: number analyzed (Participants) | 272
  Cycle1 (day 29); Post Dose | 17.19 (174)

25. Secondary Outcome: Number of Participants With Positive PD-L1 Biomarker Expression in Pre-treatment Tumor Tissue
Description: Tumor biospecimens from pre-treatment tissue samples were analyzed by immunohistochemistry for PD-L1 biomarker expression. Number of participants with positive PD-L1 biomarker expression are reported in this outcome measure.
Time Frame: At screening
Population: Biomarker analysis set for biomarkers that are measured only at screening, included all participants who received at least one dose of study drug and who had at least one screening biomarker assessment. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 397 | 407
Participants | 266 | 288

26. Secondary Outcome: PFS in PD-L1 Biomarker-Positive and PD-L1 Biomarker-Negative Subgroups
Description: PFS: time from the date of randomization to the date of the first documentation of PD according to RECIST v1.1 or death due to any cause, whichever occurred first. PFS data was censored on date of last adequate tumor assessment for participants who did not have an event (PD or death), who started new anti-cancer therapy prior to an event or for participants with an event after 2 or more missing tumor assessments. PD was defined as at least a 20% increase in the sum of all the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to relative increase of 20 %, sum must have also demonstrated an absolute > of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: as for outcome 1
Population: Biomarker positive/negative subset in FAS included participants who had at least one biomarker baseline assessment. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. "Number Analyzed" signifies number of participants evaluable for the specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 402 | 410
Months
  PD-L1 Positive Tumors: number analyzed (Participants) | 270 | 290
  PD-L1 Positive Tumors | 13.8 [11.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with event. | 7.2 [5.7 to 9.7]
  PD-L1 Negative Tumors: number analyzed (Participants) | 132 | 120
  PD-L1 Negative Tumors | 16.1 [9.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with event. | 11.1 [6.9 to 17.3]

27. Secondary Outcome: Percentage of Participants With OR in PD-L1 Biomarker-Positive and PD-L1 Biomarker-Negative Subgroups
Description: OR was defined as best overall response of CR or PR according to RECIST v1.1 as assessed by BICR recorded from date of randomization until disease progression. CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed.
Time Frame: From date of randomization until PD (maximum up to approximately 26 months)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 402 | 410
Percentage of participants
  PD-L1 Positive Tumors: number analyzed (Participants) | 270 | 290
  PD-L1 Positive Tumors | 55.2 [49.0 to 61.2] | 25.5 [20.6 to 30.9]
  PD-L1 Negative Tumors: number analyzed (Participants) | 132 | 120
  PD-L1 Negative Tumors | 47.0 [38.2 to 55.8] | 28.3 [20.5 to 37.3]

28. Secondary Outcome: Percentage of Participants With DC in Biomarker-Positive Subgroup
Description: DC was defined as a best overall response of CR, PR, or stable disease (SD) according to the RECIST v.1.1 recorded from randomization until disease progression or death due to any cause, whichever occurred first. CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed. SD was defined as PR that the sum increases by less than 20% from the nadir, (smallest sum of diameters consider baseline and all assessments prior to the time point under evaluation), but enough that a previously documented 30% decrease no longer holds.
Time Frame: From date of randomization until PD or death, whichever occurred first (maximum up to approximately 26 months)
Population: Biomarker positive subset in FAS included participants who had at least one biomarker baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 270 | 290
Percentage of participants | 84.4 [79.6 to 88.6] | 71.0 [65.4 to 76.2]

29. Secondary Outcome: TTR in Biomarker-Positive Subgroup
Description: TTR was defined as the time from randomization to the first documentation of objective tumor response (CR or PR) according to RECIST v1.1 which is subsequently confirmed. CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. All lymph nodes must decrease to normal size (short axis<10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed.
Time Frame: as for outcome 9
Population: Biomarker positive subset in FAS included participants who had at least one biomarker baseline assessment. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 149 | 74
Months | 1.6 [1.2 to 10.1] | 3.0 [1.2 to 11.6]

30. Secondary Outcome: DR in PD-L1 Biomarker-Positive and PD-L1 Biomarker-Negative Subgroups
Description: DR: time from first documentation of OR (confirmed CR or PR) to date of first documentation of PD or death due to any cause, whichever occurred first. As per RECIST version 1.1, CR: disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. PR: at least 30%< in sum of longest dimensions of target lesions taking as reference baseline sum longest dimensions. PD: defined as at least a 20% > in sum of diameters of target lesions, taking as reference the smallest sum on study (this included baseline sum if that is smallest on study). In addition to relative increase of 20%, sum must have also demonstrated an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered progression.
Time Frame: as for outcome 11
Population: as for outcome 26
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 211 | 108
Months
  PD-L1 Positive Tumors: number analyzed (Participants) | 149 | 74
  PD-L1 Positive Tumors | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of participants with event. | NA [10.9 to NA] — Median and 95% CI was not estimable due to insufficient number of participants with event.
  PD-L1 Negative Tumors: number analyzed (Participants) | 62 | 34
  PD-L1 Negative Tumors | NA [11.1 to NA] — Median and 95% CI was not estimable due to insufficient number of participants with event. | NA [9.0 to NA] — Median and 95% CI was not estimable due to insufficient number of participants with event.

31. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb) of Avelumab When Used in Combination With Axitinib
Time Frame: From start of treatment until 30 days after the end of avelumab treatment (maximum up to approximately 89 months)
Population: Immunogenicity analysis set included all participants who received at least one dose of study drug and who had at least one ADA/nAb sample collected for avelumab in "Avelumab + Axitinib" arm. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. This outcome measure was not planned to be analyzed for ''Sunitinib'' reporting group.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 433
Participants
  ADA Positive | 77
  nAb Positive | 51

32. Secondary Outcome: Time to Symptom Deterioration (TTD) for Functional Assessment of Cancer Therapy (FACT)-Kidney Symptom Index - Disease Related Symptoms (FKSI-DRS)
Description: TTD was defined as the time from date of randomization to the first time the participant's score showed a 3-point or greater decrease in FKSI-DRS. FKSI was used to assess symptoms and quality of life (QoL) for those diagnosed with advanced kidney cancer and it consisted of 19 questions. A 9-item subscale of the FKSI known as FKSI-Disease Related Symptoms subscale (FKSI-DRS). This subscale included 9 items: lack of energy, pain, losing weight, bone pain, fatigue, shortness of breath, coughing, bothered by fevers, and hematuria. Each of the 9 items was answered on a 5-point Likert-type scale ranging from 0 to 4 (0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, 4= very much). Total FKSI-DRS score = sum of the 9 item scores; total range: 0 - 36; 0 (no symptoms) to 36 (very much); higher score indicated greater presence of symptoms.
Time Frame: Date of randomization to the first time the participant's score showed a 3-point or greater decrease in FKSI-DRS (maximum up to approximately 26 months)
Population: FAS included all randomized participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Months | 4.2 [4.2 to 5.7] | 6.3 [5.5 to 8.3]

33. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQol) 5-Dimension 5 Levels (EQ-5D-5L) Utility Score
Description: EQ-5D-5L is a 5-item participant-completed questionnaire designed to assess health status in terms of a single utility score. EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Overall scores ranged from 0 to 1, with low scores representing a higher level of dysfunction. Published UK weights were used to create a single summary utility score. Utility scores range from -0.594 to 1, with higher scores representing better health status.
Time Frame: Baseline, Day 1 of Cycle 2 to Cycle 60, End of treatment (any Day from Day 1 of dosing; maximum up to approximately 89 months)
Population: FAS included all randomized participants. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Units on a scale
  Cycle 2 (Day 1): number analyzed (Participants) | 381 | 355
  Cycle 2 (Day 1) | -0.034 (0.1743) | 0.001 (0.1632)
  Cycle 3 (Day 1): number analyzed (Participants) | 356 | 317
  Cycle 3 (Day 1) | -0.023 (0.1826) | -0.017 (0.1804)
  Cycle 4 (Day 1): number analyzed (Participants) | 335 | 283
  Cycle 4 (Day 1) | -0.029 (0.1829) | -0.022 (0.1667)
  Cycle 5 (Day 1): number analyzed (Participants) | 324 | 260
  Cycle 5 (Day 1) | -0.019 (0.1622) | -0.016 (0.1826)
  Cycle 6 (Day 1): number analyzed (Participants) | 300 | 229
  Cycle 6 (Day 1) | -0.025 (0.1787) | -0.003 (0.1967)
  Cycle 7 (Day 1): number analyzed (Participants) | 276 | 202
  Cycle 7 (Day 1) | -0.018 (0.1651) | 0.008 (0.1618)
  Cycle 8 (Day 1): number analyzed (Participants) | 264 | 177
  Cycle 8 (Day 1) | -0.029 (0.1848) | 0.002 (0.1731)
  Cycle 9 (Day 1): number analyzed (Participants) | 249 | 155
  Cycle 9 (Day 1) | -0.029 (0.2021) | -0.011 (0.1662)
  Cycle 10 (Day 1): number analyzed (Participants) | 236 | 152
  Cycle 10 (Day 1) | -0.025 (0.1935) | -0.018 (0.1617)
  Cycle 11 (Day 1): number analyzed (Participants) | 228 | 138
  Cycle 11 (Day 1) | -0.020 (0.1854) | 0.004 (0.1642)
  Cycle 12 (Day 1): number analyzed (Participants) | 209 | 123
  Cycle 12 (Day 1) | -0.026 (0.1875) | -0.016 (0.1712)
  Cycle 13 (Day 1): number analyzed (Participants) | 208 | 111
  Cycle 13 (Day 1) | -0.026 (0.1777) | -0.017 (0.1549)
  Cycle 14 (Day 1): number analyzed (Participants) | 197 | 102
  Cycle 14 (Day 1) | -0.036 (0.1938) | -0.006 (0.1600)
  Cycle 15 (Day 1): number analyzed (Participants) | 192 | 102
  Cycle 15 (Day 1) | -0.036 (0.1892) | 0.018 (0.1487)
  Cycle 16 (Day 1): number analyzed (Participants) | 175 | 95
  Cycle 16 (Day 1) | -0.044 (0.1757) | 0.020 (0.1663)
  Cycle 17 (Day 1): number analyzed (Participants) | 168 | 89
  Cycle 17 (Day 1) | -0.050 (0.1950) | -0.000 (0.1675)
  Cycle 18 (Day 1): number analyzed (Participants) | 160 | 81
  Cycle 18 (Day 1) | -0.040 (0.1667) | -0.027 (0.1765)
  Cycle 19 (Day 1): number analyzed (Participants) | 148 | 78
  Cycle 19 (Day 1) | -0.059 (0.1959) | 0.003 (0.1665)
  Cycle 20 (Day 1): number analyzed (Participants) | 143 | 71
  Cycle 20 (Day 1) | -0.050 (0.1942) | 0.001 (0.1538)
  Cycle 21 (Day 1): number analyzed (Participants) | 135 | 67
  Cycle 21 (Day 1) | -0.048 (0.1902) | -0.004 (0.1904)
  Cycle 22 (Day 1): number analyzed (Participants) | 129 | 60
  Cycle 22 (Day 1) | 0.037 (0.1919) | 0.002 (0.1561)
  Cycle 23 (Day 1): number analyzed (Participants) | 118 | 58
  Cycle 23 (Day 1) | -0.033 (0.2021) | -0.028 (0.1729)
  Cycle 24 (Day 1): number analyzed (Participants) | 116 | 54
  Cycle 24 (Day 1) | -0.036 (0.1982) | 0.004 (0.1618)
  Cycle 25 (Day 1): number analyzed (Participants) | 112 | 54
  Cycle 25 (Day 1) | -0.019 (0.1825) | -0.007 (0.1678)
  Cycle 26 (Day 1): number analyzed (Participants) | 111 | 48
  Cycle 26 (Day 1) | -0.039 (0.1927) | -0.009 (0.1471)
  Cycle 27 (Day 1): number analyzed (Participants) | 107 | 45
  Cycle 27 (Day 1) | -0.046 (0.2233) | 0.014 (0.1492)
  Cycle 28 (Day 1): number analyzed (Participants) | 99 | 40
  Cycle 28 (Day 1) | -0.039 (0.2060) | -0.007 (0.1639)
  Cycle 29 (Day 1): number analyzed (Participants) | 99 | 38
  Cycle 29 (Day 1) | -0.019 (0.2095) | 0.017 (0.1601)
  Cycle 30 (Day 1): number analyzed (Participants) | 94 | 36
  Cycle 30 (Day 1) | -0.032 (0.2244) | -0.003 (0.1557)
  Cycle 31 (Day 1): number analyzed (Participants) | 90 | 35
  Cycle 31 (Day 1) | -0.042 (0.2246) | -0.009 (0.1508)
  Cycle 32 (Day 1): number analyzed (Participants) | 86 | 31
  Cycle 32 (Day 1) | -0.044 (0.2095) | 0.032 (0.1255)
  Cycle 33 (Day 1): number analyzed (Participants) | 80 | 29
  Cycle 33 (Day 1) | -0.051 (0.2294) | -0.060 (0.3550)
  Cycle 34 (Day 1): number analyzed (Participants) | 77 | 26
  Cycle 34 (Day 1) | -0.029 (0.1776) | 0.038 (0.1558)
  Cycle 35 (Day 1): number analyzed (Participants) | 66 | 26
  Cycle 35 (Day 1) | -0.010 (0.1442) | -0.002 (0.1610)
  Cycle 36 (Day 1): number analyzed (Participants) | 65 | 24
  Cycle 36 (Day 1) | -0.016 (0.1599) | 0.030 (0.1551)
  Cycle 37 (Day 1): number analyzed (Participants) | 64 | 22
  Cycle 37 (Day 1) | -0.027 (0.1507) | 0.052 (0.1601)
  Cycle 38 (Day 1): number analyzed (Participants) | 59 | 21
  Cycle 38 (Day 1) | -0.016 (0.1459) | 0.057 (0.1666)
  Cycle 39 (Day 1): number analyzed (Participants) | 56 | 18
  Cycle 39 (Day 1) | -0.042 (0.1569) | 0.052 (0.1386)
  Cycle 40 (Day 1): number analyzed (Participants) | 55 | 18
  Cycle 40 (Day 1) | -0.021 (0.1484) | 0.060 (0.1232)
  Cycle 41 (Day 1): number analyzed (Participants) | 51 | 17
  Cycle 41 (Day 1) | -0.030 (0.1492) | 0.056 (0.1853)
  Cycle 42 (Day 1): number analyzed (Participants) | 48 | 17
  Cycle 42 (Day 1) | -0.021 (0.1634) | 0.034 (0.1585)
  Cycle 43 (Day 1): number analyzed (Participants) | 45 | 16
  Cycle 43 (Day 1) | -0.031 (0.1334) | 0.011 (0.2062)
  Cycle 44 (Day 1): number analyzed (Participants) | 48 | 16
  Cycle 44 (Day 1) | -0.028 (0.1300) | 0.016 (0.2114)
  Cycle 45 (Day 1): number analyzed (Participants) | 45 | 15
  Cycle 45 (Day 1) | -0.050 (0.1442) | 0.007 (0.2191)
  Cycle 46 (Day 1): number analyzed (Participants) | 43 | 15
  Cycle 46 (Day 1) | -0.042 (0.1380) | -0.007 (0.2495)
  Cycle 47 (Day 1): number analyzed (Participants) | 39 | 13
  Cycle 47 (Day 1) | -0.019 (0.1240) | -0.015 (0.2335)
  Cycle 48 (Day 1): number analyzed (Participants) | 39 | 12
  Cycle 48 (Day 1) | -0.025 (0.1566) | 0.009 (0.2833)
  Cycle 49 (Day 1): number analyzed (Participants) | 36 | 12
  Cycle 49 (Day 1) | -0.028 (0.1356) | 0.010 (0.1873)
  Cycle 50 (Day 1): number analyzed (Participants) | 34 | 12
  Cycle 50 (Day 1) | -0.028 (0.1359) | 0.028 (0.2507)
  Cycle 51 (Day 1): number analyzed (Participants) | 26 | 11
  Cycle 51 (Day 1) | -0.011 (0.1304) | -0.010 (0.2594)
  Cycle 52 (Day 1): number analyzed (Participants) | 25 | 11
  Cycle 52 (Day 1) | -0.036 (0.1265) | -0.035 (0.2524)
  Cycle 53 (Day 1): number analyzed (Participants) | 18 | 9
  Cycle 53 (Day 1) | -0.084 (0.1437) | 0.048 (0.1308)
  Cycle 54 (Day 1): number analyzed (Participants) | 18 | 8
  Cycle 54 (Day 1) | -0.040 (0.1425) | 0.078 (0.1157)
  Cycle 55 (Day 1): number analyzed (Participants) | 14 | 5
  Cycle 55 (Day 1) | -0.046 (0.1121) | 0.051 (0.1060)
  Cycle 56 (Day 1): number analyzed (Participants) | 9 | 2
  Cycle 56 (Day 1) | -0.083 (0.1081) | 0.025 (0.1796)
  Cycle 57 (Day 1): number analyzed (Participants) | 8 | 1
  Cycle 57 (Day 1) | -0.104 (0.1347) | 0.031 (NA) — Standard deviation (SD) could not be calculated as only 1 participant was analyzed.
  Cycle 58 (Day 1): number analyzed (Participants) | 7 | 1
  Cycle 58 (Day 1) | -0.078 (0.1408) | 0.031 (NA) — SD could not be calculated as only 1 participant was analyzed.
  Cycle 59 (Day 1): number analyzed (Participants) | 5 | 0
  Cycle 59 (Day 1) | -0.106 (0.1053) |
  Cycle 60 (Day 1): number analyzed (Participants) | 3 | 0
  Cycle 60 (Day 1) | -0.040 (0.1167) |
  End of Treatment: number analyzed (Participants) | 275 | 297
  End of Treatment | -0.111 (0.2464) | -0.069 (0.2375)

34. Secondary Outcome: Change From Baseline in EQ-5D Visual Analogue Scale (VAS) Score
Description: EQ-VAS records the participant's self-rated health status from 0 (worst imaginable health status) to 100 (best imaginable health status), where higher scores indicated better health status.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Avelumab + Axitinib | Sunitinib
Number analyzed (Participants) | 442 | 444
Units on a scale
  Cycle 2 (Day 1): number analyzed (Participants) | 381 | 347
  Cycle 2 (Day 1) | -0.9 (16.12) | -0.2 (15.85)
  Cycle 3 (Day 1): number analyzed (Participants) | 355 | 312
  Cycle 3 (Day 1) | -0.4 (16.39) | 0.4 (16.44)
  Cycle 4 (Day 1): number analyzed (Participants) | 333 | 278
  Cycle 4 (Day 1) | -0.1 (17.23) | 0.7 (17.26)
  Cycle 5 (Day 1): number analyzed (Participants) | 322 | 258
  Cycle 5 (Day 1) | 0.4 (16.66) | 1.8 (16.16)
  Cycle 6 (Day 1): number analyzed (Participants) | 296 | 224
  Cycle 6 (Day 1) | 1.3 (16.05) | 2.6 (15.35)
  Cycle 7 (Day 1): number analyzed (Participants) | 275 | 197
  Cycle 7 (Day 1) | 1.2 (16.34) | 3.3 (14.91)
  Cycle 8 (Day 1): number analyzed (Participants) | 266 | 174
  Cycle 8 (Day 1) | 1.4 (16.54) | 2.9 (13.84)
  Cycle 9 (Day 1): number analyzed (Participants) | 246 | 154
  Cycle 9 (Day 1) | 2.0 (16.06) | 3.3 (13.77)
  Cycle 10 (Day 1): number analyzed (Participants) | 233 | 150
  Cycle 10 (Day 1) | 1.6 (15.12) | 2.4 (14.46)
  Cycle 11 (Day 1): number analyzed (Participants) | 225 | 135
  Cycle 11 (Day 1) | 2.5 (15.70) | 4.1 (12.91)
  Cycle 12 (Day 1): number analyzed (Participants) | 207 | 121
  Cycle 12 (Day 1) | 2.1 (14.72) | 2.6 (14.59)
  Cycle 13 (Day 1): number analyzed (Participants) | 205 | 110
  Cycle 13 (Day 1) | 3.0 (14.39) | 2.7 (14.29)
  Cycle 14 (Day 1): number analyzed (Participants) | 196 | 101
  Cycle 14 (Day 1) | 2.7 (15.07) | 3.0 (13.98)
  Cycle 15 (Day 1): number analyzed (Participants) | 192 | 101
  Cycle 15 (Day 1) | 3.1 (14.97) | 4.7 (13.63)
  Cycle 16 (Day 1): number analyzed (Participants) | 175 | 94
  Cycle 16 (Day 1) | 2.9 (15.08) | 3.6 (14.02)
  Cycle 17 (Day 1): number analyzed (Participants) | 167 | 88
  Cycle 17 (Day 1) | 3.0 (15.44) | 3.2 (12.88)
  Cycle 18 (Day 1): number analyzed (Participants) | 162 | 82
  Cycle 18 (Day 1) | 3.2 (15.31) | 2.0 (13.69)
  Cycle 19 (Day 1): number analyzed (Participants) | 147 | 78
  Cycle 19 (Day 1) | 4.5 (15.61) | 3.0 (13.10)
  Cycle 20 (Day 1): number analyzed (Participants) | 142 | 71
  Cycle 20 (Day 1) | 3.9 (15.15) | 3.1 (12.58)
  Cycle 21 (Day 1): number analyzed (Participants) | 132 | 67
  Cycle 21 (Day 1) | 3.7 (16.30) | 2.1 (13.00)
  Cycle 22 (Day 1): number analyzed (Participants) | 128 | 60
  Cycle 22 (Day 1) | 4.3 (16.43) | 2.6 (12.82)
  Cycle 23 (Day 1): number analyzed (Participants) | 117 | 58
  Cycle 23 (Day 1) | 3.7 (16.90) | 1.3 (15.16)
  Cycle 24 (Day 1): number analyzed (Participants) | 115 | 55
  Cycle 24 (Day 1) | 3.3 (18.70) | 4.5 (13.45)
  Cycle 25 (Day 1): number analyzed (Participants) | 113 | 54
  Cycle 25 (Day 1) | 4.6 (15.28) | 4.2 (14.42)
  Cycle 26 (Day 1): number analyzed (Participants) | 111 | 48
  Cycle 26 (Day 1) | 4.4 (17.10) | 3.4 (13.00)
  Cycle 27 (Day 1): number analyzed (Participants) | 106 | 45
  Cycle 27 (Day 1) | 4.7 (16.59) | 5.4 (13.43)
  Cycle 28 (Day 1): number analyzed (Participants) | 98 | 40
  Cycle 28 (Day 1) | 6.3 (16.08) | 5.0 (13.84)
  Cycle 29 (Day 1): number analyzed (Participants) | 98 | 38
  Cycle 29 (Day 1) | 4.8 (15.44) | 5.4 (14.24)
  Cycle 30 (Day 1): number analyzed (Participants) | 94 | 36
  Cycle 30 (Day 1) | 6.0 (15.78) | 5.3 (14.61)
  Cycle 31 (Day 1): number analyzed (Participants) | 89 | 35
  Cycle 31 (Day 1) | 5.7 (15.42) | 5.2 (14.88)
  Cycle 32 (Day 1): number analyzed (Participants) | 85 | 31
  Cycle 32 (Day 1) | 5.4 (16.35) | 6.0 (13.57)
  Cycle 33 (Day 1): number analyzed (Participants) | 79 | 29
  Cycle 33 (Day 1) | 5.5 (16.07) | 3.6 (20.61)
  Cycle 34 (Day 1): number analyzed (Participants) | 76 | 26
  Cycle 34 (Day 1) | 4.8 (15.25) | 6.1 (15.91)
  Cycle 35 (Day 1): number analyzed (Participants) | 65 | 26
  Cycle 35 (Day 1) | 6.0 (14.53) | 6.4 (15.61)
  Cycle 36 (Day 1): number analyzed (Participants) | 64 | 24
  Cycle 36 (Day 1) | 6.0 (15.63) | 5.2 (17.11)
  Cycle 37 (Day 1): number analyzed (Participants) | 63 | 22
  Cycle 37 (Day 1) | 5.8 (14.63) | 4.5 (15.86)
  Cycle 38 (Day 1): number analyzed (Participants) | 58 | 20
  Cycle 38 (Day 1) | 5.3 (14.58) | 4.3 (17.58)
  Cycle 39 (Day 1): number analyzed (Participants) | 56 | 18
  Cycle 39 (Day 1) | 5.3 (14.04) | 5.9 (15.75)
  Cycle 40 (Day 1): number analyzed (Participants) | 54 | 18
  Cycle 40 (Day 1) | 6.0 (15.00) | 4.7 (18.17)
  Cycle 41 (Day 1): number analyzed (Participants) | 52 | 17
  Cycle 41 (Day 1) | 5.6 (13.69) | 6.2 (18.37)
  Cycle 42 (Day 1): number analyzed (Participants) | 47 | 17
  Cycle 42 (Day 1) | 5.3 (13.68) | 5.4 (18.19)
  Cycle 43 (Day 1): number analyzed (Participants) | 44 | 16
  Cycle 43 (Day 1) | 6.6 (11.64) | 5.4 (20.14)
  Cycle 44 (Day 1): number analyzed (Participants) | 47 | 16
  Cycle 44 (Day 1) | 4.9 (13.38) | 5.1 (19.77)
  Cycle 45 (Day 1): number analyzed (Participants) | 44 | 15
  Cycle 45 (Day 1) | 6.3 (12.55) | 1.5 (17.97)
  Cycle 46 (Day 1): number analyzed (Participants) | 41 | 15
  Cycle 46 (Day 1) | 6.7 (13.25) | 0.3 (19.31)
  Cycle 47 (Day 1): number analyzed (Participants) | 38 | 13
  Cycle 47 (Day 1) | 5.4 (11.10) | 2.5 (18.07)
  Cycle 48 (Day 1): number analyzed (Participants) | 38 | 12
  Cycle 48 (Day 1) | 4.4 (11.73) | 3.5 (21.77)
  Cycle 49 (Day 1): number analyzed (Participants) | 35 | 12
  Cycle 49 (Day 1) | 4.2 (12.21) | 1.9 (21.42)
  Cycle 50 (Day 1): number analyzed (Participants) | 33 | 12
  Cycle 50 (Day 1) | 4.8 (13.07) | 2.9 (20.53)
  Cycle 51 (Day 1): number analyzed (Participants) | 26 | 10
  Cycle 51 (Day 1) | 5.8 (12.36) | 2.1 (22.93)
  Cycle 52 (Day 1): number analyzed (Participants) | 25 | 11
  Cycle 52 (Day 1) | 4.2 (11.37) | 1.5 (19.94)
  Cycle 53 (Day 1): number analyzed (Participants) | 18 | 9
  Cycle 53 (Day 1) | 3.2 (11.43) | 7.7 (16.22)
  Cycle 54 (Day 1): number analyzed (Participants) | 18 | 8
  Cycle 54 (Day 1) | 4.6 (11.54) | 7.5 (13.34)
  Cycle 55 (Day 1): number analyzed (Participants) | 14 | 5
  Cycle 55 (Day 1) | 4.6 (11.65) | 7.8 (17.89)
  Cycle 56 (Day 1): number analyzed (Participants) | 9 | 2
  Cycle 56 (Day 1) | -0.6 (8.08) | -6.0 (5.66)
  Cycle 57 (Day 1): number analyzed (Participants) | 8 | 1
  Cycle 57 (Day 1) | -1.9 (10.67) | -2.0 (NA) — SD could not be calculated as only 1 participant was analyzed.
  Cycle 58 (Day 1): number analyzed (Participants) | 7 | 1
  Cycle 58 (Day 1) | -2.1 (8.59) | -2.0 (NA) — SD could not be calculated as only 1 participant was analyzed.
  Cycle 59 (Day 1): number analyzed (Participants) | 5 | 0
  Cycle 59 (Day 1) | 0.0 (9.35) |
  Cycle 60 (Day 1): number analyzed (Participants) | 3 | 0
  Cycle 60 (Day 1) | -1.7 (16.07) |
  End of treatment: number analyzed (Participants) | 277 | 296
  End of treatment | -5.0 (19.92) | -4.3 (19.63)

ADVERSE EVENTS:
Time Frame: From start of study treatment until 90 days after last dose of study treatment (maximum up to approximately 92 months)
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. For SAEs and non-SAEs safety analysis set was used. For All-cause mortality, FAS was used.
Arm/Group | Avelumab + Axitinib | Sunitinib
All-Cause Mortality (participants affected / at risk) | 284/442 | 296/444
Serious Adverse Events (participants affected / at risk) | 231/434 | 166/439
Other Adverse Events (participants affected / at risk) | 429/434 | 433/439
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Axitinib (N=434) | Sunitinib (N=439)
Anaemia (Blood and lymphatic system disorders) | 1 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Acute coronary syndrome (Cardiac disorders) | 6 | 0
Acute myocardial infarction (Cardiac disorders) | 11 | 0
Angina pectoris (Cardiac disorders) | 3 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Autoimmune myocarditis (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 4 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial fibrosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 4 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 6 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Pituitary apoplexy (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Optic neuropathy (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 2 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 12
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 4 | 6
Asthenia (General disorders) | 4 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 6 | 0
Disease progression (General disorders) | 10 | 7
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 3 | 1
Localised oedema (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 4
Oedema peripheral (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 6
Sudden death (General disorders) | 2 | 0
Swelling (General disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 4 | 2
Cholecystitis acute (Hepatobiliary disorders) | 2 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Gallbladder rupture (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Actinomycosis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 3 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Coronavirus pneumonia (Infections and infestations) | 0 | 1
Device related bacteraemia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 6
Pneumonia aspiration (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin graft infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 5 | 3
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood corticotrophin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Myocardial necrosis marker increased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Brain hypoxia (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 5 | 4
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 1
Intracranial tumour haemorrhage (Nervous system disorders) | 0 | 1
Irregular sleep wake rhythm disorder (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1
Superficial siderosis of central nervous system (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Device breakage (Product Issues) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 9
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 5 | 6
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Renal injury (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 3
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Splinter haemorrhages (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Arterial insufficiency (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 1 | 0
Embolism venous (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 6 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Axitinib (N=434) | Sunitinib (N=439)
Anaemia (Blood and lymphatic system disorders) | 41 | 116
Leukopenia (Blood and lymphatic system disorders) | 1 | 27
Neutropenia (Blood and lymphatic system disorders) | 9 | 90
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 89
Hypothyroidism (Endocrine disorders) | 135 | 89
Abdominal pain (Gastrointestinal disorders) | 90 | 57
Abdominal pain upper (Gastrointestinal disorders) | 34 | 36
Constipation (Gastrointestinal disorders) | 97 | 73
Diarrhoea (Gastrointestinal disorders) | 303 | 228
Dry mouth (Gastrointestinal disorders) | 42 | 25
Dyspepsia (Gastrointestinal disorders) | 51 | 87
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 22 | 44
Haemorrhoids (Gastrointestinal disorders) | 21 | 31
Nausea (Gastrointestinal disorders) | 186 | 185
Oral pain (Gastrointestinal disorders) | 33 | 21
Stomatitis (Gastrointestinal disorders) | 117 | 113
Toothache (Gastrointestinal disorders) | 25 | 12
Vomiting (Gastrointestinal disorders) | 101 | 99
Asthenia (General disorders) | 83 | 83
Chest pain (General disorders) | 22 | 12
Chills (General disorders) | 75 | 38
Fatigue (General disorders) | 205 | 194
Influenza like illness (General disorders) | 34 | 22
Malaise (General disorders) | 17 | 23
Mucosal inflammation (General disorders) | 69 | 64
Oedema peripheral (General disorders) | 55 | 58
Pain (General disorders) | 22 | 23
Pyrexia (General disorders) | 74 | 65
Nasopharyngitis (Infections and infestations) | 58 | 38
Upper respiratory tract infection (Infections and infestations) | 40 | 19
Urinary tract infection (Infections and infestations) | 32 | 15
Contusion (Injury, poisoning and procedural complications) | 26 | 13
Infusion related reaction (Injury, poisoning and procedural complications) | 54 | 0
Alanine aminotransferase increased (Investigations) | 94 | 50
Amylase increased (Investigations) | 34 | 16
Aspartate aminotransferase increased (Investigations) | 83 | 59
Blood alkaline phosphatase increased (Investigations) | 21 | 24
Blood bilirubin increased (Investigations) | 22 | 20
Blood cholesterol increased (Investigations) | 23 | 16
Blood corticotrophin increased (Investigations) | 23 | 2
Blood creatine phosphokinase increased (Investigations) | 26 | 14
Blood creatinine increased (Investigations) | 64 | 37
Blood thyroid stimulating hormone increased (Investigations) | 37 | 25
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 13 | 23
Ejection fraction decreased (Investigations) | 48 | 17
Gamma-glutamyltransferase increased (Investigations) | 39 | 21
Lipase increased (Investigations) | 53 | 27
Neutrophil count decreased (Investigations) | 5 | 47
Platelet count decreased (Investigations) | 10 | 63
Weight decreased (Investigations) | 112 | 46
White blood cell count decreased (Investigations) | 4 | 38
Decreased appetite (Metabolism and nutrition disorders) | 141 | 144
Dehydration (Metabolism and nutrition disorders) | 24 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 21
Hyperkalaemia (Metabolism and nutrition disorders) | 25 | 25
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 49 | 31
Hypokalaemia (Metabolism and nutrition disorders) | 26 | 25
Hypomagnesaemia (Metabolism and nutrition disorders) | 35 | 25
Hyponatraemia (Metabolism and nutrition disorders) | 29 | 28
Hypophosphataemia (Metabolism and nutrition disorders) | 49 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 157 | 83
Back pain (Musculoskeletal and connective tissue disorders) | 118 | 80
Bone pain (Musculoskeletal and connective tissue disorders) | 23 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28 | 20
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 36 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 59 | 32
Neck pain (Musculoskeletal and connective tissue disorders) | 27 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 87 | 63
Dizziness (Nervous system disorders) | 72 | 52
Dysgeusia (Nervous system disorders) | 48 | 107
Headache (Nervous system disorders) | 122 | 85
Paraesthesia (Nervous system disorders) | 25 | 19
Taste disorder (Nervous system disorders) | 24 | 48
Anxiety (Psychiatric disorders) | 38 | 24
Insomnia (Psychiatric disorders) | 51 | 37
Haematuria (Renal and urinary disorders) | 17 | 25
Pollakiuria (Renal and urinary disorders) | 23 | 9
Proteinuria (Renal and urinary disorders) | 35 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 147 | 103
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 148 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 106 | 68
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 33 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 48 | 54
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 28 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 57 | 38
Productive cough (Respiratory, thoracic and mediastinal disorders) | 23 | 15
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 37 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 60 | 52
Erythema (Skin and subcutaneous tissue disorders) | 24 | 17
Hair colour changes (Skin and subcutaneous tissue disorders) | 2 | 29
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 160 | 162
Pruritus (Skin and subcutaneous tissue disorders) | 96 | 29
Rash (Skin and subcutaneous tissue disorders) | 74 | 54
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 29 | 11
Rash pruritic (Skin and subcutaneous tissue disorders) | 27 | 15
Skin exfoliation (Skin and subcutaneous tissue disorders) | 16 | 23
Yellow skin (Skin and subcutaneous tissue disorders) | 1 | 28
Hypertension (Vascular disorders) | 236 | 168
Hypotension (Vascular disorders) | 26 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT02684006/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT02684006/SAP_001.pdf